CLINICAL TRIAL: NCT06211062
Title: The Use of Directed Probiotics in ME/CFS: Myalgic Encephalomyelitis/Chronic Fatigue Syndrome
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Nova Southeastern University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2020-631
Record Dates: First submitted 2023-08-01; First posted 2024-01-18 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-03

CONDITIONS: ME/CFS; IBS - Irritable Bowel Syndrome
MeSH Terms: conditions — Fatigue Syndrome, Chronic; Irritable Bowel Syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double-blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Individuals with ME/CFS with IBS on active medication (Active Comparator): Individuals with ME/CFS with IBS take Floradapt Intensive GI (another name i3.1), one high dose capsule (>3x10 to the ninth power) once daily for eight weeks.
  Interventions: Drug: Floradapt Intensive GI
- Individuals with ME/CFS with IBS on placebo (Placebo Comparator): Individuals with ME/CFS with IBS take a placebo, one capsule once daily for eight weeks.
  Interventions: Other: Placebo
- Individuals with ME/CFS without IBS on active medication (Active Comparator): Individuals with ME/CFS without IBS take Floradapt Intensive GI (another name i3.1), one high dose capsule (>3x10 to the ninth power) once daily for eight weeks.
  Interventions: Drug: Floradapt Intensive GI
- Individuals with ME/CFS without IBS on placebo (Placebo Comparator): Individuals with ME/CFS without IBS take a placebo, one capsule once daily for eight weeks.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Floradapt Intensive GI — one capsule daily for the eight week intervention
  Other Names: i3.1
  Arms: Individuals with ME/CFS with IBS on active medication; Individuals with ME/CFS without IBS on active medication
Other: Placebo — one capsule daily for the eight week intervention
  Arms: Individuals with ME/CFS with IBS on placebo; Individuals with ME/CFS without IBS on placebo

SUMMARY:
This clinical study aims to evaluate the use of i3.1 probiotic in participants who meet the Institute of Medicine (Canadian Consensus Criteria) case definition for ME/CFS and who may or may not be diagnosed with irritable bowel syndrome (IBS). The main questions it aims to answer are:

* how effective is the usage of the i3.1 probiotic to reduce gastrointestinal (GI) inflammation and normalize the GI and systemic/brain interface?
* how well is it working on IBS severity? The study sample is 100 male and female participants aged 45 to 70 years with ME/CFS (per the Canadian Consensus Criteria); one-half of the participants will have co-morbid IBS (per Rome IV criteria). Participants will receive an i3.1 or a placebo and be assessed at baseline, at eight weeks, and at 12 weeks (four weeks post-treatment completion).

DETAILED DESCRIPTION:
This single-site comparison study will be performed on 100 participants, 45 to 70 years of age, who meet the Institute of Medicine (Canadian Consensus Criteria) case definition for ME/CFS and who may or may not be diagnosed with the irritable bowel syndrome (IBS), according to the Rome IV criteria. In this study, we will evaluate using the i3.1 probiotic compared to placebo. This is a randomized, placebo-controlled trial with four study arms that will include 25 participants per arm: Individuals with ME/CFS with and without IBS, who will take either the active medication i3.1 or placebo.

ELIGIBILITY:
Inclusion Criteria: eligible if all of the following apply:

* Meets IOM ME/CFS case definition criteria,
* Co-morbid IBS: meets RomeIV criteria for alternating or diarrhea-predominant IBS as reported during screening (technically diagnosed by a physician),
* Able to provide consent to study,
* Patients of childbearing potential must practice effective contraception during the study and be willing to continue contraception for at least six months after the intervention,
* agrees to participate in online surveys and follow-up visits.

Exclusion Criteria: ineligible if any of the following apply:

* Probiotics in the past eight weeks,
* Antibiotics in the past eight weeks,
* Pregnancy or lactating women,
* Medical conditions including short bowel syndrome, celiac disease, biliary disease, pancreatitis, inflammatory bowel disease (Crohn's disease, ulcerative colitis), severe cardiovascular, neurological condition, or liver failure,
* Gastrointestinal surgery within six months of study entry,
* History of psychiatric disorder, alcohol or illicit drug abuse.

Ages: 45 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-12-20 (Actual); Primary Completion 2026-02-24 (Estimated); Study Completion 2026-02-24 (Estimated)

PRIMARY OUTCOMES:
The Incidence of Intervention-Related Adverse Events [Safety] | from baseline to the eight week visit
  Safety will be assessed by documenting the frequency and severity of adverse events using a standardized form at each visit.
The Measurement of Biomarker Response to an Intervention in the Blood [Efficacy] | from baseline to the eight week visit
  The inflammation biomarkers panel will be measured at baseline and during the eight-week visit.
  Inflammation biomarkers analyses (such as zonulin, LPS (lipopolysaccharide) endotoxin, LBP (lipopolysaccharide-binding protein)
level of CRP (C-reactive protein) | from baseline to the eight week visit
  CRP (C-reactive protein) will be measured at baseline and the eight-week visit (The Measurement of Biomarker Response)
The pro-inflammatory cytokines level e.g. IL-1, IL-6, and TNF-α | from baseline to the eight week visit
  The Measurement of Biomarker Response : cytokine panel.
The Symptom Severity Measurement [Efficacy] | from baseline to the eight week visit
  The symptom severity will be measured as a change of scores on the DePaul Symptom Questionnaire (DSQ) from baseline to eight-week visit. The severity and frequency are calculated on the Likert scale, where for severity 0 refers to symptoms not present, and 4 is for very severe, and for the frequency: 0 is for none of the time, and 4 is for all of the time. The score range is from 0 to 216. A higher score means a worse outcome (symptoms are present more often with more severity).

SECONDARY OUTCOMES:
The Impact on the Irritable Bowel Syndrome (IBS) Severity | from baseline to the eight week
  The impact on the Irritable Bowel Syndrome (IBS) severity will be assessed by response to intervention based on the change in score on the IBS-SSS (Irritable Bowel Syndrome Symptom Severity Scale) questionnaire from a baseline visit to an eight-week visit. Scores response on a 100-point visual analogue scale range from 0 to 500. Subjects can be categorized as mild (75-175), moderate (175-300), or severe (>300) IBS. A decrease of 50 points is associated with a clinically meaningful improvement.
The IBS-related Quality of Life Measurement | from the eight week visit to the 12 week visit
  The measurement will be provided using the IBS-QOL (the Irritable Bowel Syndrome Quality of Life Measurement) questionnaire every visit from baseline to week eight. Each item is related on the Likert scale, ranging from 1 to 5 (1 as "not at all", 5 as "extremely"). Total score ranges from 34 to 170; higher scores mean a lower life quality. A decrease of 10 points is a clinically meaningful improvement.

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Klimas, MD, Principal Investigator — Nova Southeastern University, Institute for Neuroimmune Medicine
Locations (1):
- Institute for Neuroimmune Medicine, Fort Lauderdale, Florida, United States

IPD SHARING:
Plan to Share IPD: No
No plan available